CLINICAL TRIAL: NCT04698837
Title: AeroCOVID 1: Understanding Potential Airborne Transmission and the Protective Value of Type II Surgical Masks in SARS-CoV-2 Using Patient Proximity Environmental Sampling With a Highly Efficient Bioaerosol and Droplet Collection Dummy
Brief Title: Understanding Potential Airborne Transmission and the Protective Value of Type II Surgical Masks in SARS-CoV-2
Acronym: aeroCOVID1
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Lucerne University of Applied Sciences and Arts (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-02768
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: SARS-CoV-2
Keywords: Airborne transmission; Aerosol transmission; Surgical masks

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Modes of transmission of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and specifically the proportion of airborne transmission in this infection is unknown. In the aeroCOVID study, a highly efficient bioaerosol and droplet sampling dummy is used to emulate a susceptible healthcare worker (HCW) and to perform patient proximity sampling. The dummy will measure the dummy-inhaled dose of SARS-CoV-2 in two particle size fractions in a standardized interaction with hospitalized coronavirus disease 2019 (COVID-19) patients. All measurements are performed in a masked and unmasked dummy setup in parallel, in order to gain further information on the protection of type II masks against the respective particle size exposure.

DETAILED DESCRIPTION:
Modes of interpersonal transmission in SARS-CoV-2 are to date only incompletely understood and require further investigation in order to define best preventive measures. Although a dichotomization of inhaled particles by particle size is an oversimplification and a large particle size does not exclude shortterm airborne behavior, the suspension time of virus containing particles and the probability of particles to accumulate in room air is primarily defined by particle size distribution. Particles with a size below 10 µm have a high probability of accumulation due to their mean suspension time of minutes to hours.

The study aims to measure the total amount of virus copies per particle size fraction inhaled by a highly efficient sampling dummy emulating a susceptible HCW in a standardized interaction with hospitalized COVID-19 patients. As a secondary endpoint, the proportion of culturable virus in each setup is measured as well.

Sampling is done in using two parallel bioaerosol and droplet sampling dummies - one type II masked and one with an unmasked dummy head as inlet - in order to gain additional information on the protective effect of type II surgical masks in a real-life exhaled particle size distribution in hospitalized COVID patients. The sampling dummy consists of a real size face relief connected to an 60° inlet cone, a cyclone for collection of particles >10 µm and a laminar flow water-based condensation bioaerosol collector for particle collection below 10 µm particle size.

After patient proximity sampling, a nasopharyngeal swab for SARS-CoV-2 polymerase chain reaction (PCR) assay is performed. Relevant indoor climate parameters like temperature, humidity and carbon dioxide (CO2) as well as room characteristics as air change rate are recorded as well.

ELIGIBILITY:
Inclusion Criteria:

* positive SARS-CoV-2 PCR or antigen test from a nasopharyngeal or oropharyngeal swab
* ≥18 years of age
* ability to give consent
* ability to follow simple instructions

Exclusion Criteria:

* symptom onset more than 10 days prior to inclusion
* pregnancy
* lack of written informed consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is performed with hospitalized COVID-19 patients at Inselspital, Bern University hospital. The study site hospital is a tertiary university hospital treating COVID-19 patients on normal hospital wards as well as in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Total amount of dummy-inhaled virus copies per 30 minutes sampling per size fraction (>10 µm, <10 µm) | 30 minutes sampling

SECONDARY OUTCOMES:
Viability of dummy-inhaled viable virus per size fraction (>10 µm, and <10 µm) | 30 minutes sampling
Reduction of dummy-inhaled virus copies per 30 minutes sampling in a type II-masked setup, as compared to unmasked, per size fraction (>10 µm, <10 µm) | 30 minutes sampling

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Jent, MD, Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland